CLINICAL TRIAL: NCT05509517
Title: Remote Heart Rhythm Monitoring Using Photoplethysmography-based Smartphone Technology for the Early Detection of Atrial Fibrillation and Adverse Events After Cardiac Surgery
Brief Title: A Clinical Trial of the Use of Remote Heart Rhythm Monitoring With a Smartphone After Cardiac Surgery
Acronym: SURGICAL-AF 2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: S64572
Record Dates: First submitted 2022-07-12; First posted 2022-08-22 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2022-11

CONDITIONS: Atrial Fibrillation and Flutter; Atrial Fibrillation; Postoperative Complications; Arrhythmia
Keywords: Atrial Fibrillation; Digital Health; Artificial Intelligence; Cardiac Surgery; Postoperative atrial fibrillation (POAF)
MeSH Terms: conditions — Atrial Fibrillation; Postoperative Complications; Arrhythmias, Cardiac

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rhythm monitoring group (Experimental): Patients randomized to the rhythm monitoring arm will assess their heart rhythm with a photoplethismography (PPG) based smartphone application (FibriCheck™). Measurements are performed three times daily and while experiencing symptoms. The patients start measuring immediately after discharge and continues until the scheduled postoperative consultation with the cardiologist or cardiac surgeon at 21-91days after discharge.
  Interventions: Diagnostic Test: Photoplethysmography based smartphone application for heart rhythm analysis (FibriCheck™)
- Usual care (No Intervention): Patients randomized to the rhythm monitoring arm will be discharged without protocol mandated rhythm monitoring. A postoperative consultation is scheduled with the cardiologist or cardiac surgeon at 21-91days after discharge.

INTERVENTIONS:
Diagnostic Test: Photoplethysmography based smartphone application for heart rhythm analysis (FibriCheck™) — Heart Rhythm assessment using the FibriCheck™ application with the patient's proprietary smartphone, three times daily, from discharge until follow-up consultation (day 21-91 after discharge).
  Arms: Rhythm monitoring group

SUMMARY:
The objective of the study is to evaluate the clinical consequences following the detection of postoperative atrial fibrillation or flutter (POAF) using a remote heart rhythm monitoring strategy with a photoplethysmography based smartphone technology in the early postoperative period after discharge.

DETAILED DESCRIPTION:
A predefined subgroup analysis of the outcomes described below will be performed in the following subgroups:

* Subjects not on anticoagulation drug therapy (for a planned duration of >45 days) at discharge.
* Subjects with no history of AF prior to surgery and no POAF lasting >24h in hospital.
* Subjects with a CHADSVASC score ≥ 4 or a CHADSVASC score ≥ 2 with at least one additional risk factor associated with the risk of developing POAF.

additional risk factors include:

* chronic obstructive pulmonary disease
* sleep apnea
* impaired renal function
* left atrial enlargement
* elevated body mass index
* combined CABG with valve repair or replacement

ELIGIBILITY:
Inclusion Criteria:

* Subject underwent any of (including a combination of) the following surgical procedures during index hospitalization. (coronary artery bypass graft, surgical repair or replacement of a cardiac valve)
* Subject provides informed consent
* Subject understands and agrees to comply with planned study procedures.
* Subject is able to perform heart rhythm measurement using the FibriCheck application at home.

Exclusion Criteria:

* Pacemaker dependent heart rhythm
* Permanent AF/Aflutter or AF/Aflutter present at the time of inclusion
* Insufficient cognitive or comprehensive level of Dutch to participate to the trial.
* No smartphone available at home.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Actual)
Dates: Start 2021-11-02 (Actual); Primary Completion 2023-07-05 (Actual); Study Completion 2023-09-04 (Actual)

PRIMARY OUTCOMES:
Proportion of participants with any of the following therapeutic interventions (composite 4-point endpoint) | 91 days
  Any of the following therapeutic interventions:
  * Initiation or unplanned continuation of anticoagulation drug therapy resulting from arrhythmia detection
  * Initiation or increase in dose regimen of anti-arrhythmic drug therapy (Vaughan-williams class 1 or 3)
  * Cardioversion
  * Cardiac implantable electronic device (CIED) implantation
Time to detection of a postoperative adverse event | 91 days
  Prespecified postoperative adverse events:
  1.1. Acute respiratory insufficiency 1.2. Pleural effusion 1.3. Pneumonia 1.4. Pulmonary Embolism 1.5. Pneumothorax 1.6. Atelectasis, leading to respiratory insufficiency
  2.1. Acute myocardial infarction 2.2. Symptomatic arrhythmia 2.3. Pericardial effusion 2.4. Pericarditis 2.5. Endocarditis 2.6. Systemic embolism 2.7. Cardiogenic shock
  3.1. Acute stoke including cerebrovascular accident (CVA) and transient ischemic attack (TIA)
  4.1. Renal failure, defined as: >50% increase in serum creatinine or initiation of renal replacement therapy 4.2. Urinary tract infection, requiring antibiotic treatment
  5. Wound related complications requiring surgical intervention or antibiotic treatment.
  6. Sepsis
  7. Other unplanned hospitalisations will be classified by the research team as 'postoperative adverse event' or 'unrelated to the cardiac surgery procedure'. Such events will be reported with the study results.

SECONDARY OUTCOMES:
Time to primary endpoint (primary outcome 1) | 91 days
Proportion of participants with initiation or unplanned continuation of anticoagulation drug therapy resulting from arrhythmia detection | 91 days
Post-operative atrial fibrillation (POAF) detection rate | 91 days
Time to POAF detection | 91 days
POAF detection rate in subjects with an indication for anticoagulation | 91 days
Detection rate of POAF lasting more than 6 hours | 91 days
The EQ-5D-5L questionnaire score evolution between inclusion and follow-up consultation | 91 days
  EQ-5D-5L is a EuroQol five-dimension scale questionnaire. The participant rates his or her own level of impairment across dimensions (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression) from 1 to 5 and global health rating on a visual analogue scale (EQ-VAS) from 1 to 100.
Number of mayor adverse cardiac outcomes (All-cause death, Ischemic stroke, Myocardial infarction, Systemic embolism) | Two years
  Hierarchical secondary outcomes (will be analysed if the primary outcome is positive)
Number of mayor adverse cardiac outcomes (secondary outcome 9) with addition of cardiovascular hospitalisations | Two years
  Hierarchical secondary outcomes (will be analysed if the primary outcome is positive)

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospitals Leuven, Leuven, Belgium